CLINICAL TRIAL: NCT00733096
Title: A 3-arm Multi-center, Randomized Controlled Study Comparing Transforaminal Corticosteroid, Transforaminal Etanercept and Transforaminal Saline for Lumbosacral Radiculopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency); National Naval Medical Center (U.S. Federal Agency); Womack Army Medical Center (U.S. Federal Agency); Landstuhl Regional Medical Center (U.S. Federal Agency); Massachusetts General Hospital (Other)
Responsible Party: Steven P. cohen, Walter Reed Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-6891
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2010-09

CONDITIONS: Lumbosacral Radiculopathy
Keywords: radiculopathy; sciatica; low back pain
MeSH Terms: conditions — Radiculopathy; Sciatica; Low Back Pain | interventions — Etanercept; Methylprednisolone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Epidural etanercept 4 mg, two doses 2 weeks apart
  Interventions: Drug: etanercept
- 2 (Active Comparator): Epidural methylprednisolone 60 mg, two doses 2 weeks apart
  Interventions: Drug: methylprednisolone
- 3 (Placebo Comparator): Epidural saline, two doses 2 weeks apart
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: etanercept — Two transforaminal epidural injections of 4 mg, two weeks apart
  Arms: 1
Drug: methylprednisolone — Two transforaminal epidural steroid injections with 60 mg, two weeks apart
  Arms: 2
Drug: normal saline — Two transforaminal epidural saline injections, two weeks apart
  Arms: 3

SUMMARY:
Lumbosacral radiculopathy is one of the leading of cause of disability in the U.S. and worldwide. Among recent reviews evaluating epidural steroid injections, some 1 but not all 2 concluded them to be effective in the long-term. In our own double-blind, placebo-controlled study evaluating epidural etanercept, the results showed significant benefit in favor of the etanercept group, but no subject was included with a duration of pain > 9 months, and the results of this study have yet to be replicated.

Currently, epidural steroid injections are the most frequently performed procedures in pain clinics across the U.S. However, epidural steroids may benefit only a select group of patients. The literature on treating sciatica is notable for a lack of randomized comparative studies involving various treatments. The objective of this project is to conduct a 3-arm study to determine the efficacy of 1) transforaminal epidural corticosteroids; and 2) transforaminal epidural etanercept, in patients with lumbosacral radiculopathy.

DETAILED DESCRIPTION:
This is a 3-arm multi-center, randomized, double-blind, placebo-controlled study comparing two treatments with transforaminal epidural saline. Each group will receive a 2nd procedure identical to the first 2 weeks after the initial procedure.

Seventy-eight study participants will be randomized via a computerized randomization system using SPSS software in groups of 6 at each institution by a research nurse not involved in patient care. There will be 26 patients in each of the 3 groups. A physician unaware of the patient's treatment group will place 22-gauge needles in the relevant foramen under fluoroscopic guidance as determined by patient's symptoms and MRI findings. Once correct placement is confirmed by contrast injection, the blinded physician will leave the room and another physician will inject the medication. In group I, this will be 60 mg of depo-methylprednisolone. In group II, this will be 4 mg of etanercept reconstituted in 2 ml of sterile water. In group III, this will be normal saline.

Two weeks after the initial procedure, an identical procedure to the first one will be done by the same physician or his designate. In addition to the study medication, each patient in each group will receive 0.5 ml of 0.5% bupivacaine local anesthetic for immediate pain relief during both injections before the study drug is delivered. The efficacy of blinding will be assessed by a disinterested observer unaware of the randomization results after the second procedure before discharge. Follow-up visits will be conducted one, three and six months after the second injection, for those subjects who continue to experience > 50% pain relief.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic low back pain of radicular origin of > 4 weeks but < 6 months duration.
2. Leg pain > back pain.
3. Failure of conservative therapy to include physical and pharmacotherapy.
4. MRI evidence of a lateral or paracentral herniated disc corresponding to the patient's radicular symptoms.

Exclusion Criteria:

1. Uncontrolled coagulopathy.
2. Pregnancy, which will be ruled out by a urine pregnancy test in women of childbearing age.
3. Allergy to contrast dye or amide local anesthetics.
4. Previous epidural steroid injection within last year.
5. Unstable medical or psychiatric condition (e.g. unstable angina, congestive heart failure or severe depression) that could preclude an optimal treatment response.
6. Rheumatoid arthritis or spondylarthropathy.
7. Unstable neurological condition (e.g. multiple sclerosis)
8. Systemic infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Womack Army Medical Center, Fort Bragg, North Carolina

REFERENCES:
- [Background] Mulleman D, Mammou S, Griffoul I, Watier H, Goupille P. Pathophysiology of disk-related sciatica. I.--Evidence supporting a chemical component. Joint Bone Spine. 2006 Mar;73(2):151-8. doi: 10.1016/j.jbspin.2005.03.003. Epub 2005 Jun 22. PMID 16046173
- [Derived] Cohen SP, White RL, Kurihara C, Larkin TM, Chang A, Griffith SR, Gilligan C, Larkin R, Morlando B, Pasquina PF, Yaksh TL, Nguyen C. Epidural steroids, etanercept, or saline in subacute sciatica: a multicenter, randomized trial. Ann Intern Med. 2012 Apr 17;156(8):551-9. doi: 10.7326/0003-4819-156-8-201204170-00397. PMID 22508732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 patients were enrolled between 2008 and 2011
Pre-assignment Details: 80 patients were excluded before assignment
Groups:
- Steroid: Two epidural steroid injections
- Etanercept: Two epidural etanercept injections
- Saline: Two epidural saline injections
Period: Overall Study
Arm/Group | Steroid | Etanercept | Saline
Started | 28 | 26 | 30
Completed | 28 | 26 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid | Etanercept | Saline | Total
Number analyzed (Participants) | 28 | 26 | 30 | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.7) | 43.2 (8.9) | 42.3 (10.7) | 42.29 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 11 | 25
  Male | 22 | 18 | 19 | 59
Region of Enrollment [Number; unit: participants]
  United States | 28 | 26 | 30 | 84

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Leg Pain Score
Description: 0-10 pain score. 0= no pain, 10= worst imaginable pain.
Time Frame: 1 month
Population: Patients who received epidural steroid injections
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Steroid | Etanercept | Saline
Number analyzed (Participants) | 28 | 26 | 30
units on a scale | 2.54 [1.36 to 3.69] | 3.56 [2.35 to 4.72] | 3.78 [2.72 to 4.85]

2. Secondary Outcome: Oswestry Disability Score
Description: 0-100%. 0= no disability, 100% is complete disability
Time Frame: 1 month
Population: Patients who received epidural steroid injections
Measure: Mean (95% Confidence Interval); unit: percentage of disability out of 100%
Arm/Group | Steroid | Etanercept | Saline
Number analyzed (Participants) | 28 | 26 | 30
percentage of disability out of 100% | 22.4 [16.64 to 31.55] | 40.26 [32.91 to 47.61] | 30.00 [23.2 to 36.69]

3. Secondary Outcome: Global Perceived Effect
Description: Satisfaction. Number of participants with positive perceived global satisfaction.
Time Frame: 1 month
Population: Subjects who underwent epidural steroid injections
Measure: Number; unit: participants
Arm/Group | Steroid | Etanercept | Saline
Number analyzed (Participants) | 28 | 26 | 30
participants | 23 | 15 | 17

4. Secondary Outcome: Medication Reduction
Description: Number of people who reduced medications
Time Frame: 1 month
Population: Patients who underwent epidural steroid injections
Measure: Number; unit: participants
Arm/Group | Steroid | Etanercept | Saline
Number analyzed (Participants) | 28 | 26 | 30
participants | 17 | 9 | 14

ADVERSE EVENTS:
Arm/Group | Steroid | Etanercept | Saline
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26 | 0/30
Other Adverse Events (participants affected / at risk) | 1/28 | 5/26 | 6/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Steroid (N=28) | Etanercept (N=26) | Saline (N=30)
Worsening pain (General disorders) | 0 | 4 | 3
Nonlocal infection (Infections and infestations) | 0 | 1 | 3
Nonlocal rash (Infections and infestations) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Subjects who failed to obtain benefit were unblinded after 1-month, which limits conclusions regarding long-term efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No